CLINICAL TRIAL: NCT04246931
Title: Evaluation of Perception and Knowledge of Adherence to COPD Inhalation Therapy at Patient, GP and Pulmonologist Level
Brief Title: Adherence Evaluation in COPD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chiesi SA/NV (Other)
Responsible Party: Sponsor
Other Study IDs: Chiesi_NIS_0003
Record Dates: First submitted 2020-01-15; First posted 2020-01-29 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Adherence, Treatment; COPD
MeSH Terms: conditions — Treatment Adherence and Compliance; Pulmonary Disease, Chronic Obstructive | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pulmonologists: Interviews with pulmonologists
  Interventions: Other: No intervention (survey)
- General practitioners: Interviews with general practitioners
  Interventions: Other: No intervention (survey)
- Patients: Survey with COPD patients
  Interventions: Other: No intervention (survey)

INTERVENTIONS:
Other: No intervention (survey) — No intervention -> survey at 1 timepoint

SUMMARY:
The rationale of this study is to have a better understanding of the perception of the pulmonologists, general practitioners and patients of adherence (causes, main consequences, supportive tools,..) and the use of TAI-questionnaire (appreciation, usability,…) by interviewing pulmonologists & general practitioners and a survey with patients. Based on the outcome, projects and tools can be developed to help health care professionals to motivate patients to improve adherence and to help patients to increase their adherence to inhalation therapy.

ELIGIBILITY:
Inclusion Criteria:

Pulmonologists or general practitioners or COPD patient (suffering from COPD treated with inhalation therapy)

Exclusion Criteria:

Not applicable

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Pulmonologists, general practicioners and COPD patients
Sampling Method: Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-03-15 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Knowledge and perception of adherence | Baseline
  Gathering knowledge based on semi-structured interview (definition, causes, consequences of bad adherence,...)

SECONDARY OUTCOMES:
Test of the adherence to inhalers-questionnaire (TAI) | Baseline
  Evaluate the usability of 'Test of the adherence to inhalers'-questionnaire (TAI) based on semi-structured interview

CONTACTS AND LOCATIONS:
Overall Officials: Sofie Geelissen, PhD, Study Chair — Chiesi Belgium
Locations (1):
- Medistrat, Lasne, Belgium

IPD SHARING:
Plan to Share IPD: Undecided